CLINICAL TRIAL: NCT06281418
Title: Postoperative Pain Management Following Laparoscopic Cholecystectomy- Intraperitoneal Granisetron
Brief Title: Postoperative Intraperitoneal Pain Management Following Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Hoda Mohamed, Teaching Assistant- Pharmacy Practice & Clinical Pharmacy, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5-24
Record Dates: First submitted 2024-02-18; First posted 2024-02-28 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain
Keywords: laparoscopic; post-operative pain; serotonin 5HT3 receptor antagonist
MeSH Terms: conditions — Pain, Postoperative | interventions — Granisetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Placebo Comparator): 2 ml IP normal saline (0.9 % NaCl)
  Interventions: Other: Normal saline
- Intervention arm (Experimental): 2ml IP granisetron (1 mg/mL)
  Interventions: Drug: Granisetron 1 Mg/mL Intravenous Solution

INTERVENTIONS:
Drug: Granisetron 1 Mg/mL Intravenous Solution — 2mL intraperitoneal adminstration of granisetron (1 mg/mL)
  Arms: Intervention arm
Other: Normal saline — 2 ml IP normal saline (0.9% NaCl)
  Arms: Control arm

SUMMARY:
Postoperative pain management is essential and the inability to treat acute pain appropriately in the first 48 postoperative hours represents a risk factor for developing chronic pain. No. study has investigated IP granisetron as an adjuvant to standard care for postoperative pain management in patients undergoing LC.

DETAILED DESCRIPTION:
Postoperative pain is a main challenge for delayed hospital discharge in Laparoscopic cholecystectomy. . Postoperative pain management is essential and the inability to treat acute pain appropriately in the first 48 postoperative hours represents a risk factor for developing chronic pain. Granisetron is frequently used as a premedication to avoid postoperative nausea and vomiting in patients who have undergone general anesthesia. The purpose of this study is evaluating the efficacy and tolerability of IP granisetron on postoperative pain control in patients undergoing LC

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo elective LC.
* Adults (males and/or females) between the ages of 18-70 years old.

Exclusion Criteria:

* Chronic pain other than cholelithiasis.
* Patients who received analgesics or sedatives 24 h before scheduled surgery.
* Severe hepatic (Child Pugh Class B and C) and renal dysfunction (CrCl <30ml/min)
* Previous allergic response to granisetron.
* Pregnancy and lactation
* Patients with communication problems, cognitive dysfunction, or psychological disorders
* Daily corticosteroid use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
VAS score | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours
  Pain intensity: VAS score

SECONDARY OUTCOMES:
Time to analgesic request | 24 hours
  Time to first rescue analgesic request
Quality of life (QoL) after laparoscopic cholecystectomy (LC) | 3 months
  Gastrointestinal Quality of Life Index questionnaire for QOL assessment with calculation of the score; most desirable option: 4 points, least desirable option: 0 points and GIQLI score: sum of the point. GIQLI ranges from 0 to 80 with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hepatology and Tropical Research Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bayoumi HM, Abdelaziz DH, Boraii S, Bendas ER, El Said NO. Intraperitoneal Granisetron for Post-Laparoscopic Cholecystectomy Pain Management: A Double-Blinded, Randomized Controlled Trial. Pharmacotherapy. 2025 Sep;45(9):547-556. doi: 10.1002/phar.70046. Epub 2025 Jul 23. PMID 40698525